CLINICAL TRIAL: NCT05021679
Title: Activity and Mobility Promotion (AMP): Implementation and Impact of a Multifaceted Intervention to Increase Mobility in Hospital Patients
Brief Title: AMP Step Wedge Trial
Acronym: AMP SWT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB00270215
Record Dates: First submitted 2021-08-16; First posted 2021-08-25 (Actual); Last update posted 2024-04-25 (Actual); Status verified 2024-04

CONDITIONS: Immobility; Disability
Keywords: Activity; Mobility; Hospital-acquired disability
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Intervention Model Description: Step-wedge clinical trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- AMP Implementation (Experimental)
  Interventions: Other: AMP Implementation

INTERVENTIONS:
Other: AMP Implementation — Each study site will implement the Johns Hopkins AMP program at different times. The AMP program includes nursing staff training on the goals of AMP, how to complete mobility-focused outcome measures, set mobility goals, and to safely mobilize/ambulate patients. The AMP program also includes embedding these outcome measures and mobility goals into electronic medical records and producing weekly/monthly reports that show how often nursing staff score patient mobility and help patients meet daily activity goals.

SUMMARY:
Annually, more than 35 million patients are hospitalized in the United States. Many of these will experience hospital-acquired loss of physical functioning due to a lack of mobility during their in-patient stay. Such loss includes difficulties performing basic activities, such as rising from a chair, toileting, or ambulating. This loss of function may increase hospital length of stay (LOS), nursing home placement, and decrease mobility and participation in community activities even years after hospitalization. Prevention of this hospital-acquired functional loss is critical. Even the sickest hospitalized patients (e.g., those in the intensive care unit [ICU]), can safely and feasibly benefit from early mobilization. In the non-ICU setting there is evidence that patient mobilization reduces LOS and hospital costs, while improving patient satisfaction and physical and psychological outcomes. The overall objective of this proposed project is to evaluate the implementation and impact of a transdisciplinary and multifaceted mobility program (Johns Hopkins Activity and Mobility Promotion - AMP) on clinical outcomes among hospitalized adults. In addition to clinical outcomes, we will identify barriers and facilitators to high-performance program adoption. Results of this project will provide critical new insights on the effectiveness of AMP and inform dissemination and implementation nationwide.

ELIGIBILITY:
Inclusion Criteria:

* All adult patients admitted to study hospital unit
* Analysis will only include those with lengths of stay >=3 days

Exclusion Criteria:

* Patients with active do-not-resuscitate (DNR) order
* <18 years old

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16676 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2024-04-01 (Actual); Study Completion 2024-04-01 (Actual)

PRIMARY OUTCOMES:
% of patients meeting daily mobility goal | 39 months
  Mobility goal is set and measured using the Johns Hopkins Highest Level of Mobility (JH-HLM) Scale
% of patients with mobility measurements documented daily | 39 months
  Mobility documentation to include Activity Measure for Post-Acute Care (AM-PAC) and JH-HLM
% of patients receiving physical and/or occupational therapy consults | 39 months
  To be extracted from electronic medical record

SECONDARY OUTCOMES:
Hospital length of stay (days) | 39 months
  To be extracted from electronic medical record
Discharge disposition status | 39 months
  Count of where patients are discharged to (e.g,. home, inpatient rehab unit) assessed by extraction from electronic medical record.
Number of physical and occupational therapy visits received during inpatient stay | 39 months
  To be extracted from electronic medical record
Number of hospital-acquired morbidities | 39 months
  Includes falls, pressure injury, and venous thromboembolism. To be extracted from electronic medical record
Number of patients with 30-day readmissions | 39 months
  To be extracted from electronic medical record
Employee injuries resulting from patient mobilization | 39 months
  Number of employee injuries from facilitating patient mobility as assessed by medical record extraction

CONTACTS AND LOCATIONS:
Overall Officials: Sapna Kudchadkar, MD, Principal Investigator — Johns Hopkins University; Erik Hoyer, PhD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins Hospital, Baltimore, Maryland, United States